CLINICAL TRIAL: NCT05577104
Title: The Comparison of Negative Pressure Wound Therapy (NPWT) and Conventional Moist Dressings in the Wound Bed Preparation for Diabetic Foot Ulcers
Brief Title: Wound Bed Preparation for Diabetic Foot Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, YinWu, attending doctor of Department of Burn and Plastic Surgery,Nanjing First Hospital, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20220825-08
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Diabetic Foot
Keywords: diabetic foot ulcers; negative pressure wound therapy; wound blood perfusion; neutrophil extracellular traps
MeSH Terms: conditions — Diabetic Foot | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: The patients with diabetic foot ulcers (DFUs)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the NPWT group (Experimental): For patients in the NPWT group, the wound bed preparation was facilitated by VAC device.
  Interventions: Procedure: Negative pressure wound therapy (NPWT)
- the control group (Active Comparator): For patients in the control group, the wound bed preparation was facilitated by alginates dressing change method.
  Interventions: Procedure: conventional moist dressings

INTERVENTIONS:
Procedure: Negative pressure wound therapy (NPWT) — For patients in the NPWT group, the wound bed preparation was facilitated by vacuum-assisted closure (VAC).
  Arms: the NPWT group
Procedure: conventional moist dressings — For patients in the control group, the wound bed preparation was facilitated by conventional dressing change method (with alginates ).
  Arms: the control group

SUMMARY:
The study objective was to compare the efficacy of NPWT versus alginates dressings on the wound bed preparation prior to STSG surgery, as well as investigating the underlying mechanisms.

DETAILED DESCRIPTION:
The diabetic foot ulcers (DFUs) are major complications of patients with diabetes mellitus. Split thickness skin graft (STSG) surgery is a cost-effective method for the rapid healing of DFUs. The aim of this study was to compare the efficacy of negative pressure wound therapy (NPWT) using vacuum-assisted closure (VAC) device versus conventional moist dressings (alginates) on the wound bed preparation prior to STSG surgery for patients with chronic DFUs.

This ia a prospective, randomized controlled trial. All the patients were randomly divided into two groups: the NPWT group or the control group. Once the DFUs wound was filled with healthy granulation tissues, STSG surgery was performed. The primary endpoint included the time to STSG surgery (the duration from first surgical debridement to STSG surgery). The secondary endpoints included the survival rates of skin graft, the wound blood perfusion, the wound neutrophil extracellular traps (NETs) formation, and polarization of M1 or M2 macrophages in the DFUs wounds of the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with DFUs aged 20-80 years.
2. Wagner grade 2 to 3.
3. Chronic DFUs wounds (duration of disease ≥ 2 weeks).
4. Ankle brachial ratio (ABI) 0.5～0.9, wound area 8~20 cm2.

Exclusion Criteria:

1. Patients who were unable to complete the follow-up were not included,
2. Pregnant or nursing mothers were not included.
3. Patients with foot ulcers other than diabetes, peripheral vascular disease, organ dysfunctions (heart failure, respiratory failure, liver dysfunction, renal impairment or intestinal failure), or autoimmune diseases (rheumatoid arthritis, ankylosing spondylitis, systemic lupus erythematosus, Sjogren's syndrome, connective tissues disease or systemic vasculitis) were not included.
4. Patients who received growth factors or hyperbaric oxygen therapies for the DFUs wounds within one month were not included.
5. Patients who had medications (such as corticosteroids, immunosuppressive agents or chemotherapy) within six months were not included.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-10 (Estimated)

PRIMARY OUTCOMES:
the time to STSG surgery | 3 months post debridement
  the duration from first surgical debridement to STSG surgery

SECONDARY OUTCOMES:
the wound blood perfusion | Before the radical surgical debridement (Day 0), After NPWT or conventional dressing change therapy for 6 days (Day 6).
  The blood perfusion of the DFUs wounds were evaluated by the laser speckle contrast imaging (LSCI) instrument. The higher value means a better outcome.
the wound neutrophil extracellular traps (NETs) formation | Before the radical surgical debridement (Day 0), After NPWT or conventional dressing change therapy for 6 days (Day 6).
  The wound granulation tissues (1 mL) were collected from the DFU wound of patients. The wound granulation tissues were stained for NETs by immunofluorescence. Samples were stained with anti-human neutrophil elastase antibody and anti-human myeloperoxidase antibody. Visualization was performed with confocal microscopy. The higher number of NETs means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Yin Wu, phD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
The Study Protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF), Clinical Study Report (CSR) are to be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will become available on December,2023. The data will become available for 1 year.
Access Criteria: everyone
URL: http://www.stats.gov.cn/tjsj/

REFERENCES:
- [Result] Tettelbach W, Cazzell S, Sigal F, Caporusso JM, Agnew PS, Hanft J, Dove C. A multicentre prospective randomised controlled comparative parallel study of dehydrated human umbilical cord (EpiCord) allograft for the treatment of diabetic foot ulcers. Int Wound J. 2019 Feb;16(1):122-130. doi: 10.1111/iwj.13001. Epub 2018 Sep 24. PMID 30246926
- See also: Pubmed — https://pubmed.ncbi.nlm.nih.gov/30246926/